CLINICAL TRIAL: NCT01994499
Title: Randomized Study Comparing Pleural Drainage by Videothoracoscopy to Medical Drainage in Infectious Pleural Effusion
Acronym: VIDMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/009/HP
Record Dates: First submitted 2013-10-30; First posted 2013-11-25 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Infectious Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- videothoracoscopy drainage (Experimental): videothoracoscopy drainage of pleural effusion
  Interventions: Device: Videothoracoscopy drainage
- Medical pleural drainage (Active Comparator): Medical drainage
  Interventions: Drug: Medical drainage

INTERVENTIONS:
Device: Videothoracoscopy drainage — videothoracoscopy drainage of pleural effusion
  Arms: videothoracoscopy drainage
Drug: Medical drainage — Medical pleural drainage
  Arms: Medical pleural drainage

SUMMARY:
Infectious pleural effusion is a classic complication of pneumonia and often require pleural drainage.

There is no consensus between surgical drainage and medical drainage indication in first intention to treat an empyema.

Usually surgery is proposed in second intention after failure of medical drainage.

Videothoracoscopy is well accepted in diagnosis and treatment of pleural pathologies. The morbidity of this approach is very low with good results and become the gold standard in different pleural diseases. The medical drainage can be also very efficient but its results depends of the evolution of the pleural effusion. The rate of failure is estimated around 25%.

Then, the aim of our study is to compare surgical drainage and medical drainage in first intention. The first end-point will be the hospital stay (day). Hospital discharge will be strict, following different objective criteria of healing allowing comparison between these two approaches of drainage.

To answer this question we will randomized 50 patients in 2 years with a multicenter recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Infectious pleural effusion diagnosed by pleural punction with biologic features of infection: C Reactive Protein level >5 mg/L, White cells counts > 10000 G/L, Temperature >38°c, effusion with a ph<7,2 or presence of polynuclear, and radiologic features of effusion requiring drainage (>1/5 thoracic volume)

Exclusion Criteria:

* prior thoracic surgery, past history of pleural effusion
* compressive effusion which should be treated in emergency
* Pregnancy
* No acceptance of the protocol by the informed patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Hospital Stay in days | patients will be followed for the duration of the hopital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jean-marc baste, MD, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - University Hospital, Amiens
  - University Hospital, Caen
  - UH Rouen, Rouen